CLINICAL TRIAL: NCT06765616
Title: Adebrelimab Injection (PD-L1) Combined With Short Course Radiotherapy and Chemotherapy for Neoadjuvant Therapy of Locally Advanced Rectal Cancer: a Multicenter, Single Arm Prospective Study
Brief Title: Adebrelimab Injection (PD-L1) Combined With Short Course Radiotherapy and Chemotherapy for Neoadjuvant Therapy of Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Feng Tian (Other Government)
Responsible Party: Sponsor-Investigator, Feng Tian, Dr, Shandong Provincial Hospital
Organization: Shandong Provincial Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-OBU-SD-CRC-II-004
Record Dates: First submitted 2024-12-22; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Rectal Cancer; Advanced Stage Colorectal Cancer; Radiotherapy
Keywords: Immune checkpoint inhibitors；Adebrelimab Injection
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab Injection combined with radiotherapy and chemotherapy (Experimental): Radiotherapy regimen: SCRT short-term radiotherapy of 5 × 5Gy Immunotherapy regimen: Adebrelimab Injection 1200 mg or 20 mg/kg, iv., followed by administration on the 1st day of each subsequent chemotherapy cycle.
  Chemotherapy regimen: CAPOX regimen (chemotherapy cycle d1, to chemotherapy cycle d14):
  Oxaliplatin 130 mg/m2 iv d1
  Capecitabine 1000 mg/m2 po bid d1~14
  Repeat every 3 weeks for 6 cycles
  After completing 6 cycles of chemotherapy, the patient underwent TME surgery 2-3 weeks later.
  Interventions: Drug: Adebrelimab Injection combined with radiotherapy and chemotherapy

INTERVENTIONS:
Drug: Adebrelimab Injection combined with radiotherapy and chemotherapy — Radiotherapy regimen: SCRT short-term radiotherapy of 5 × 5Gy Immunotherapy regimen: Adebrelimab Injection 1200 mg or 20 mg/kg, iv., followed by administration on the 1st day of each subsequent chemotherapy cycle.
  Chemotherapy regimen: CAPOX regimen (chemotherapy cycle d1, to chemotherapy cycle d14):
  Oxaliplatin 130 mg/m2 iv d1
  Capecitabine 1000 mg/m2 po bid d1~14
  Repeat every 3 weeks for 6 cycles
  After completing 6 cycles of chemotherapy, the patient underwent TME surgery 2-3 weeks later.

SUMMARY:
This study is a multicenter, single arm, prospective study aimed at evaluating the efficacy and safety of adebelimab combined with short course radiotherapy (5 * 5Gy) and chemotherapy as preoperative neoadjuvant therapy for locally advanced rectal cancer patients. In the study, all subjects who met the inclusion criteria will receive a combination of adebelimab, short course radiotherapy (5 * 5Gy), and CAPOX chemotherapy as neoadjuvant therapy according to the study plan. TME surgery will be performed 2-3 weeks after the last dose of neoadjuvant therapy. If the surgery cannot be performed within the time window specified in the protocol (such as delayed adverse reactions, etc.), the researcher will consider the actual clinical situation of the subjects comprehensively.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent before implementing any experimental procedures;
2. Male or female, aged 18 or above and 85 or below;
3. Patients diagnosed with rectal adenocarcinoma through primary lesion biopsy and histopathological examination;
4. Patients with cT stage ≥ T3 or cN stage N1+, M0 or EMVI (+) or MRF (+) or suspected lateral lymph node metastasis (>5mm) who are determined to be operable and require neoadjuvant therapy through imaging and colonoscopy examination.
5. According to imaging and colonoscopy examination, the main body of the patient's tumor is located ≤ 15cm away from the anal edge;
6. According to the criteria for evaluating the efficacy of solid tumors (RECIST version 1.1), there should be at least one measurable lesion on imaging;
7. The patient has not received any anti-tumor treatment in the past, including but not limited to surgery, radiotherapy, chemotherapy, immunotherapy, targeted therapy, etc;
8. ECOG score 0-1 points;
9. Adequate organ function, subjects must meet the following laboratory indicators:

   * In the past 14 days without using granulocyte colony-stimulating factor, the absolute neutrophil count (ANC) was ≥ 1.5x109/L.
   * Platelets ≥ 100 × 109/L without blood transfusion in the past 14 days.
   * Hemoglobin>9g/dL in the past 14 days without blood transfusion or use of erythropoietin;
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN);
   * Aspartate transaminase (AST) and alanine transaminase (ALT) levels are ≤ 2.5 × ULN
   * Blood creatinine ≤ 1.5 × ULN and creatinine clearance rate (calculated using Cockcroft Gault formula) ≥ 60 ml/min;
   * Good coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN;
   * Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
   * The myocardial enzyme spectrum is within the normal range (simple laboratory abnormalities that are deemed clinically insignificant by the researchers are also allowed to be included)
10. For female subjects of childbearing age, a urine or serum pregnancy test with negative results should be conducted within 3 days prior to the first administration of the study drug (Day 1 of the first cycle). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Non childbearing women are defined as those who have been postmenopausal for at least one year or have undergone surgical sterilization or hysterectomy; If there is a risk of conception, all subjects (male or female) must use contraceptive measures with an annual failure rate of less than 1% throughout the entire treatment period until 120 days after the last administration of the study drug (or 180 days after the last administration of chemotherapy drug).

Exclusion Criteria:

1. Patients diagnosed with other malignant tumors that have not been cured within 5 years before the first administration (excluding skin basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ that has undergone radical resection);
2. Late stage rectal cancer patients with distant metastasis;
3. Currently participating in interventional clinical research treatment, or having received other research drugs or used research instruments for treatment within 4 weeks before the first administration;
4. Previously received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs, or drugs that stimulate or synergistically inhibit T cell receptors (such as CTLA-4, OX-40, CD137);
5. Have received systemic treatment of traditional Chinese patent medicines and simple preparations with anti-tumor indications or drugs with immunomodulatory effect within 2 weeks before the first administration;
6. Within 2 years prior to the first administration, there has been an active autoimmune disease requiring systemic treatment (such as the use of disease relieving drugs, corticosteroids, or immunosuppressants). Alternative therapies (such as thyroid hormone, insulin, or physiological glucocorticoids used for adrenal or pituitary insufficiency) are not considered systemic treatments;
7. Within 7 days prior to the first administration of the study, the individual was receiving systemic corticosteroid therapy (excluding topical corticosteroids via nasal spray, inhalation, or other routes) or any other form of immunosuppressive therapy;Note: Physiological doses of glucocorticoids (≤ 10 mg/day of prednisone or equivalent) are allowed to be used;
8. Known allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
9. Those who are known to be allergic to the active ingredients or excipients of the investigational drug Adabelimab and combination chemotherapy drugs;
10. Prior to commencing treatment, the individual has not fully recovered from any toxicity and/or complications caused by any intervention measures (i.e., ≤ grade 1 or baseline, excluding fatigue or hair loss);
11. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
12. Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected is greater than the upper limit of normal value in the laboratory of the research center);Note: hepatitis B patients who meet the following criteria can also be included in the group:

    * Prior to the first administration, if the HBV viral load is less than 1000 copies/ml (200 IU/ml), subjects should receive anti HBV treatment throughout the entire study chemotherapy period to avoid viral reactivation
    * For subjects with anti HBc (+), HBsAg (-), anti HBs (-), and HBV viral load (-), prophylactic anti HBV treatment is not necessary, but close monitoring of viral reactivation is necessary
13. Active HCV infected subjects (HCV antibody positive and HCV-RNA level above the detection limit);
14. Administer a live vaccine within 30 days prior to the first dose (Day 1 of the first cycle);Note: It is allowed to receive inactivated vaccine for seasonal influenza within 30 days before the first administration; However, intranasal administration of attenuated live influenza vaccine is not allowed.
15. Pregnant or lactating women;
16. There are any serious or uncontrollable systemic diseases, such as:

    * Resting electrocardiogram shows significant and difficult to control abnormalities in rhythm, conduction, or morphology, such as complete left bundle branch block, grade II or higher heart block, ventricular arrhythmia, or atrial fibrillation;
    * Unstable angina pectoris, congestive heart failure, chronic heart failure classified as NYHA ≥ 2;
    * Myocardial infarction occurred within 6 months prior to enrollment;
    * Poor blood pressure control (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg);
    * A history of non infectious pneumonia requiring corticosteroid treatment within the year prior to the first administration, or current clinical active interstitial lung disease;
    * Active pulmonary tuberculosis;
    * There are active or uncontrolled infections that require systemic treatment;
    * There is clinical active diverticulitis, abdominal abscess, and gastrointestinal obstruction;
    * Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
    * Poor control of diabetes (FBG>10mmol/L);
    * Urine routine shows urinary protein ≥++and confirms 24-hour urinary protein quantification>1.0 g;
    * Patients with mental disorders who are unable to cooperate with treatment;
17. Medical history or disease evidence, abnormal treatment or laboratory test values that may interfere with the trial results, hinder the full participation of the subjects in the study, or other situations that the researchers believe are not suitable for inclusion. The researchers believe that there are other potential risks and they are not suitable to participate in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission rate (pCR) | From enrollment to the end of surgery,assessed up to 6 months
  Pathological complete remission rate (pCR)

SECONDARY OUTCOMES:
Objective response rate (ORR) | The evaluation time from enrollment to the first efficacy evaluation is up to 3 months
  Objective response rate (ORR)
Major Pathological Response Rate (MPR) | From enrollment to the end of surgery,assessed up to 6 months
  Major Pathological Response Rate (MPR)
R0 resection rate | From enrollment to the end of surgery,assessed up to 6 months
  R0 resection rate
Adverse reaction incidence rate | From enrollment to 90 days after the last medication
  Adverse reaction incidence rate

CONTACTS AND LOCATIONS:
Overall Officials: Changqing Jing, Professor, Study Director — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No